CLINICAL TRIAL: NCT03136783
Title: New Tumor Models in Three Dimensions and in a Human Skin Environment for Personalized Melanoma Therapy
Acronym: SkinTher
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0021
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Melanoma (Skin)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with stage IV melanoma (Other)
  Interventions: Other: Development of the most specific physiologically relevant experimental patient models

INTERVENTIONS:
Other: Development of the most specific physiologically relevant experimental patient models — Development of the most specific physiologically relevant experimental patient models: organotypic culture of biopsies, reconstituted skin (equivalents of dermis with melanoma, dermis equivalents and epidermis with melanoma), and in vitro evaluation The response of tumor cells to different combinations of targeted therapy molecules

SUMMARY:
The choice of treatment of patients with metastatic melanoma depends on the status of B-RAF of the tumor: in the absence of mutation, treatment with immunotherapy (currently anti-PD1) is proposed in the first line; When B-RAF is mutated, treatment with targeted therapies is retained: B-RAF and MEK inhibitors are prescribed in combination (vemurafenib + cobimetinib or dabrafenib + trametinib).

Patient response rates for targeted therapies range from 50 to 60%, and the occurrence of sometimes severe side effects is not predictable. There are currently no predictive biomarkers of patients' response to targeted therapy molecules. The in vitro evaluation of the intrinsic sensitivity of the cells of patients to different combinations of targeted therapy molecules would make it possible to propose the best therapeutic combinations. The cutaneous metastases are chosen in the model because of easy access to collect tumor tissue.

The most relevant in vitro models for mimicking cutaneous melanoma metastases are explant cultures and human skin equivalents.

ELIGIBILITY:
Inclusion Criteria:

* Major Patients,
* patients with melanoma (stage IV) with cutaneous metastases,
* seronegative HIV, HBV, HCV, HTLV1.

Exclusion Criteria:

* Absence of cutaneous metastasis or in transit
* HIV or HBV or HCV or HTLV1 seropositivity
* Patient minor, patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-09-22 (Estimated); Study Completion 2019-09-22 (Estimated)

PRIMARY OUTCOMES:
Evaluating in vitro the response of tumor cells to different combinations of targeted therapy molecules | 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France